CLINICAL TRIAL: NCT04670718
Title: The Use of a Novel Optical Coherence Tomography (OCT) Probe in Assessment of Endoscopic and Surgical Resection Specimen of Gastrointestinal Tract
Brief Title: The Use of a OCT Probe in Assessment of Endoscopic and Surgical Resection Specimen of Gastrointestinal Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Associate Consultant, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020.570
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Gastrointestinal neoplasm; Optical coherence tomography
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OCT probe (Experimental): The examination of gastrointestinal tract resected specimen with the use of the OCT probe
  Interventions: Device: Optical Coherence Tomography Probe

INTERVENTIONS:
Device: Optical Coherence Tomography Probe — Use of OCT probe for examination of gastrointestinal tract

SUMMARY:
This is a pilot study aiming to investigate the ability of a novel Optical Coherence Tomography (OCT) probe in assessing the different layers of the gastrointestinal tract and the depth of invasion of early neoplasia, utilising surgically and endoscopically resected specimens

DETAILED DESCRIPTION:
Endoscopic treatment of early neoplasia in the gastrointestinal tract has been established as the standard therapy in the past decade. Various endoscopic resection techniques have been developed, such as endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD), to ensure complete removal of such lesions and avoid recurrence. Successful endoscopic resection of early gastrointestinal (GI) neoplasia relies on accurate pre-procedural prediction of the margin and depth of invasion of the corresponding lesions. Generally, GI neoplasia (even carcinoma) confined to the mucosa layer could be safely removed endoscopically with margin negative resection and minimal chance of lymph node involvement.

Image-enhanced endoscopy or endoscopic ultrasonography has been used as the modality of pre-resection assessment on the depth of invasion. Chromoendoscopy and digital enhancement such as magnifying Narrow Band Imaging (NBI) focus on characterization of the surface morphology and the vascular structures and predict the depth of invasion instead of direct depth measurement. Endoscopic ultrasonography allows good visualization of the different layers of GI tract, but the ability to differentiate early mucosal (T1a) or submucosal invasive (T1b) cancer remains limited owing to its low resolution (>100um). A small proportion of patients subjected for endoscopic resection had invasive cancer not curable by endoscopic means and require additional surgery afterwards. There is thus a potential role for further refinement of imaging technique to allow better prediction of tumor depth in early GI neoplasia.

Optical coherence tomography (OCT) is a novel high spatial-resolution, cross-sectional imaging technique that allows visualization of biological tissue at higher resolution (~10um). It has been used routinely in the field of ophthalmology for retinal assessment. Earlier studies have also confirmed the potential application in the gastrointestinal tract with a probe-based design to be placed within an endoscopy.

The Department of Mechanical and Automation Engineering from the Chinese University of Hong Kong have recently designed a novel OCT probe that could be placed within the working channel of an endoscope. In-vitro experiment with porcine intestinal model demonstrated its ability to provide high-resolution images with visualization of different layers of the GI tract. The investigators therefore design this pilot study to assess the application of the OCT probe in human resected tissue specimen to assess the ability in determining different layers of GI tract and depth of invasion of GI tumors.

The current pilot study is designed aiming to assess the ability of the novel OCT probe in visualization of the layers of the human GI tract and depth of invasion of GI neoplasia in resected surgical and endoscopic specimens. There would be two parts of the study:

1. To visualize normal gastrointestinal tract in a resected surgical specimen of esophageal, stomach, small bowel and colonic tissue.
2. To assess the depth of invasion of the neoplastic tissue in surgical specimens as well as endoscopic (ESD) specimens

ELIGIBILITY:
Inclusion Criteria:

1. Patients with esophageal, gastric or colonic cancer undergoing elective surgical resection
2. Patients with early esophageal, gastric or colonic neoplasia undergoing endoscopic resection (Endoscopic submucosal dissection)

Exclusion Criteria:

* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Visualisation of gastrointestinal tract | 1 day
  Visualisation of different layers of gastrointestinal tract. Ability to differentiate mucosa and submucosa and muscular propria layer. (Yes or No).

SECONDARY OUTCOMES:
Ability to asses depth of invasion of resected GI early tumor | 1 day
  Ability to assess depth of invasion of resected GI early tumor

CONTACTS AND LOCATIONS:
Overall Officials: Hon Chi Yip, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong